CLINICAL TRIAL: NCT02401191
Title: A Non-controlled, Open Study for Assessing the Safety and Effectiveness of a Twice-daily FEX 60 mg - PE 10 mg (FEX60/PE10) Fixed Combination Tablet in Patients With Allergic Rhinitis
Brief Title: A Study Assessing the Safety and Effectiveness of FEX60/PE10 Fixed Combination Tablet in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEXHYL07477
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEX60/PE10 (Experimental): Internal use of FEX60/PE10 combination tablet will be administered twice daily (1 tablet per intake) for 2 weeks
  Interventions: Drug: FEX60/PE10

INTERVENTIONS:
Drug: FEX60/PE10 — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To assess the safety of twice-daily fexofenadine 60 mg/phenylephrine 10 mg (FEX60/PE10) combination tablet in patients with allergic rhinitis.

Secondary Objective:

To evaluate the effectiveness of a twice-daily FEX60/PE10 combination tablet on nasal symptoms (sneezing, rhinorrhea, and nasal congestion), and daily activity impairment.

DETAILED DESCRIPTION:
It will be 22 days at minimum and up to 32 days depending on screening, treatment, and post-treatment observation allowances.

ELIGIBILITY:
Inclusion criteria:

* Outpatients with a history of seasonal or perennial allergic rhinitis for at least 1 year confirmed by positive skin prick test to out or indoor allergens (wheal ≥3mm compared to control [diluent]) or positive specific IgE Antibody test (ie, radioallergosorbent test [RAST], etc.) on the day of provisional inclusion in the trial.
* Patients who meet the following criteria of symptom score. (The symptom score is rated according to the 'Severity of nasal symptoms'):

  1. Nasal congestion score is consistently from 2 to 3 but not 4 for the last 3 days of the screening period.
  2. Score of sneezing or rhinorrhea is consistently 2 or 3 but not 4 throughout the last 3 days of the screening period.
* Patients aged 15 years or older, with no restriction on gender.
* Patients written informed consent.
* Females with childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of study drug and adequate contraception during the study.

Exclusion criteria:

* Patients with nasal diseases (hypertrophic rhinitis, paranasal sinusitis, nasal polyps, acute rhinitis, deviation of the nasal septum, etc.) that could interfere with judgment of the efficacy of the investigational product (IP) and patients developing cold-like symptoms during screening period.
* Patients with severe asthma, bronchiectasis, severe hepatic, renal, or cardiac dysfunction, hematological, endocrine disease, and other serious complications.
* Patients with unstable medical conditions like diabetes mellitus, heart failure, hepatic and renal impairment.
* Patients with a history of epilepsy or with organic brain disease, which may cause epilepsy.
* Patients who have taken any of the following medications that may affect the evaluation of the IP, Patients using intranasal or systemic decongestants if they are not stopped 3 days before the inclusion visit.

  1. Within 1 week prior to the day of registration:

     * Intranasal or oral:

       * Antiallergic drugs, antihistamines, anticholinergic agents, vasoconstrictor, antihistamine-containing cold remedies, agents that can be expected to have an antiallergic/antihistaminic effect (including Chinese medicines and glycyrrhizin), and other agents that are indicated for allergic symptoms (sneezing, rhinorrhea, nasal congestion, etc.).
     * Agents that may affect the blood concentration of Fexofenadine (FEX) (macrolide antibiotics, azole fungicides, and preparations containing aluminum hydroxide/magnesium hydroxide).
  2. Within 2 weeks prior to the day of registration:

     o Steroids, immunosuppressant, and nonspecific alternative therapy (histamine-containing gamma-globulin preparations etc).
  3. Within 4 weeks prior to the day of registration:

     * Patients receiving oral, nasal, inhaled corticosteroids.
     * Depot steroid preparations.
* Patients using sodium cromoglycate/nedocromil or leukotriene modifiers if they are not stopped 14 days before the inclusion.
* Patients under immunotherapy if specific immunotherapy has been started or dose changed approximately 1 month preceding enrolment in the study, (doses should maintain the same dose throughout the trial).
* Patients suffering from Upper Respiratory Tract Infection, sinusitis or acute otitis media within 30 days before the inclusion visit.
* Patients who are participating in another study or who have previously participated in another study within the previous 6 months prior to the day of registration.
* Patients who are considered by the Investigator/sub-investigator to be unsuitable for enrolment in the study for any other criterion or previously participated in this study.
* Patients with a history of hypersensitivity to antihistamines or antiallergic agents including FEX.
* Patients with severe hypertension or severe coronary artery disease, narrow angle glaucoma, urinary retention, or those who have shown sensitivity to adrenergic agents (manifestations include insomnia dizziness, weakness, tremor, or arrhythmias).
* Patients receiving monoamine oxidase (MAO) inhibitor therapy or within 2 weeks prior to the day of registration.
* Women who are pregnant, possibly pregnant, or breast-feeding.
* Patients with underlying hepatobiliary disease. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (Solicited AE reporting) | From intake of FEX60/PE10 up to approximately 2 weeks
Changes from baseline in the nasal congestion score based on the patient's symptom diary | After 2 weeks treatment

SECONDARY OUTCOMES:
Change from baseline in the total score of 3 nasal symptoms (sneezing, rhinorrhea, and nasal congestion) | After 2 weeks treatment
Change in the total score of 3 nasal symptoms on a daily basis | After 2 weeks treatment
Change in the total score of 3 nasal symptoms during daytime | After 2 weeks treatment
Change in the total score of 3 nasal symptoms during night-time | After 2 weeks treatment
Change in the daily activity impairment score | After 2 weeks treatment
Change in the daily activity impairment score on a daily basis | After 2 weeks treatment
Change in the daily activity impairment score during daytime | After 2 weeks treatment
Change in the daily activity impairment score during night-time | After 2 weeks treatment
Change in nasal findings from baseline: color of inferior turbinate mucosa | After 2 weeks treatment
Change in nasal findings from baseline: congestion of inferior turbinate mucosa | After 2 weeks treatment
Change in nasal findings from baseline: consistency of discharge | After 2 weeks treatment
Assessment of patient's impression after treatment based on patient's symptom diary | After 2 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi Administrative Office, Tokyo, Japan